CLINICAL TRIAL: NCT07101146
Title: Pathological Myopia and Quality of Life: An Exploratory Study of Patient Outcomes and Perceptions
Brief Title: 100 High Myopia Patient-reported Outcomes (PRO) and Performance Outcomes (PERFO)
Acronym: PPO100
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P22-06
Record Dates: First submitted 2025-07-24; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: High Myopia

STUDY DESIGN:
Intervention Model Description: Prospective, longitudinal, interventional, exploratory, non-randomized, single-center study including patients with pathological myopia
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Qualitative Phase (Other): The "Qualitative" phase, estimated to last six months, will be conducted on a panel of up to 30 patients with hight myopia for the purpose of conducting semi-structured interviews and pre-tests to calibrate the Perf Outcome parameters.
  Interventions: Other: Quality of life questionnaire; Other: Performance Outcomes (PerfO); Other: Semi-structured interviews
- Exploratory Phase (Other): The "Exploratory" phase, estimated to last 18 months, will be conducted on a panel of 70 patients with hight myopia in order to explore the validity of Perf Outcome.
  Interventions: Other: Quality of life questionnaire; Other: Performance Outcomes (PerfO)

INTERVENTIONS:
Other: Quality of life questionnaire — The NEI-RQL-42 (National Eye Institute Refractive Quality of Life) questionnaire will be self-administered via a secure online platform to assess the impact of pathological myopia on quality of life.
Other: Performance Outcomes (PerfO) — Three tests are planned to assess the impact of high myopia on critical aspects of mobility and safety, with the possibility of adjusting their scope based on pilot data.
  * The first test involves an assessment of driving on a simulator, designed to evaluate the performance of detecting pedestrians in peripheral vision, with and without glare.
  * The second test focuses on assessing mobility and obstacle avoidance under six levels of brightness.
  * The third test evaluates visual search ability. It consists of finding spheres in everyday scenes in an apartment with six levels of contrast tested.
Other: Semi-structured interviews — Semi-structured interviews will only be offered to patients recruited in Phase 1 Qualitative and aim to further explore the information gathered from the NEI-RQL-42 questionnaire responses and the difficulties encountered during the performance tasks in the laboratory, by exploring in more detail the limitations encountered by patients with pathological myopia in their daily activities. These interviews will help identify the specific causes of the difficulties encountered, as well as the environmental conditions that may create discomfort or increased hardship.
  Arms: Qualitative Phase

SUMMARY:
Prospective, longitudinal, interventional, exploratory, non-randomized, single-center study including patients with pathological myopia .

DETAILED DESCRIPTION:
This project will be conducted in two phases, with a qualitative study and an exploratory phase.

There is a clinical need to better understand the progression of myopic complications with diffuse choroidal atrophy (DCA Cat. 2) and choroidal patch atrophy (CPA Cat. 3) and their impact on everyday life.

The first phase is a qualitative study whose objectives are

1. to study the parameters (ceiling and floor effects) and assess the reliability of performance tasks in relation to perceived difficulties,
2. to use interviews to gather information on the difficulties reported in everyday life, the causes, and the environmental conditions leading to a reduction in activity in a population of myopic patients with retinal complications.

The second phase will consist of a quantitative exploratory pilot study aimed at comparing the performance of diffuse choroidal atrophy (DCA) and choroidal patch atrophy (CPA) patients in order to highlight any differences between the two in tasks involving mobility and obstacle avoidance, visual search, and driving

ELIGIBILITY:
Inclusion Criteria:

Patients with pathological myopia and diffuse choroidal atrophy (DCA, Cat. 2 Meta PM)

* Age ≥ 18 years and ≤ 55 years;
* Patient consenting to be included in the study;
* Examination and follow-up in at least one of the participating centers;
* Severe pathological myopia with an axial length ≥ 26.5 mm in both eyes;
* Presence of diffuse atrophy (category 2 of the Meta-PM classification) in the better eye;
* Affiliated with or covered by a social security system.

Pathological myopic patients with patch choroidal atrophy (PCA,

Cat. 3 Meta PM):

* Age ≥ 18 years and ≤ 55 years;
* Patients who consent to be included in the study;
* Examination and follow-up at least one of the participating centers;
* High myopia with an axial length ≥ 26.5 mm in both eyes;
* Presence of patch atrophy (category 3 of the Meta-PM classification) in the better eye;
* Affiliated with or beneficiary of a social security system.

Exclusion Criteria:

* Identified genetic syndromic myopia, including Stickler syndromes type 1 and 2 (collagen 2A1 and 11A1), Marfan syndrome (fibrillin), Ehler-Danlos syndrome type 4 (lysyl-protocollagen hydroxylase), and Knobloch syndrome (collagen 18A).
* Patient unwilling to participate or be followed up at one of the participating centers.
* Binocular visual acuity ≥ 1 logMar (<0.1 on the decimal scale).
* Media opacities preventing quality imaging, including cataracts.
* Patients benefiting from legal protection measures.
* Pregnant or breastfeeding women.
* Individuals who may not be able to tolerate the driving simulator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Simulator driving test:Evaluation of pedestrian detection performance using peripheral vision | 2 months
  This test aims to evaluate drivers' performance in detecting pedestrians in their peripheral vision,with and without glare.
  Participants' performance will be measured in terms of speed and accuracy in detecting pedestrians.
Locomotion assessment | 2 months
  This task aims to measure visual abilities to move safely in an environment where the participant finds their way and avoids obstacles present in the course.
  Performance is measured by walking speed and the accuracy of foot positioning.
Visual search in VR | 2 months
  Score calculated based on the total number of targets identified in two minutes and the number of mistakes made.

CONTACTS AND LOCATIONS:
Overall Officials: Elise PHILIPPAKIS, MD, Principal Investigator — Hôpital Fondation Adolphe de Rothschild